CLINICAL TRIAL: NCT04651920
Title: A Study on Association Between Homologous Recombination Genes and the Homologous Recombination Deficiency Status in Chinese Population With Epithelial Ovarian Cancer
Brief Title: A Study on Association Between HR Genes and the HRD Status in Chinese Epithelial Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-HRD2
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-03

CONDITIONS: Epithelial Ovarian Cancer; Chinese; Homologous Recombination Deficiency; BRCA1 Mutation; BRCA2 Mutation; Prognosis; Homologous Recombination Genes
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — All patients accept evaluation of homologous recombination deficiency model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epithelial ovarian cancer patients sensitive to platinum based chemotherapy
  Interventions: Genetic: Evaluation of homologous recombination deficiency score
- Epithelial ovarian cancer patients resistant to platinum based chemotherapy
  Interventions: Genetic: Evaluation of homologous recombination deficiency score

INTERVENTIONS:
Genetic: Evaluation of homologous recombination deficiency score — Evaluation of homologous recombination deficiency score which is based on the loss of heterozygosity (LOH), telomere allele imbalance (TAI) and large-scale state transitions (LST)

SUMMARY:
The association between homologous recombination (HR) gene mutations and homologous recombination deficiency (HRD) status in Chinese epithelial ovarian cancer (EOC) patients is little known. This study would recruit 400 Chinese EOC patients with known targeted gene mutations via a multi-panel testing of 27 genes, including BRCA1/BRCA2. All patients accept evaluation of HRD model, which is based on the loss of heterozygosity (LOH), telomere allele imbalance (TAI) and large-scale state transitions (LST). The mutated genes, HRD score model and their relationship with the prognosis, would provide a full description of for the Chinese EOC patients, and a potential explanation of platinum-resistance in such population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Pathological confirmation of epithelial ovarian cancer
* With available tumor tissues
* Given consents to participate the study

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Chinese population with confirmed diagnosis of epithelial ovarian cancer with known targeted gene mutations via a multi-panel testing of 27 genes and known resistance to platinum-based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Homologous recombination deficiency (HRD) score | Two years
  The HRD score for individual patient is a scale describing her HRD status. The score model is calculated by the analysis for three types of important molecular mechanism: loss of heterozygosity (LOH), telomere allele imbalance (TAI) and large-scale state transitions (LST). The minimum value is 0, but the maximun value is not available. Higher scores mean more sensitivity to poly-ADP-ribose polymerase inhibitor.

SECONDARY OUTCOMES:
Progression-free survival | Five years
  Progression-free survival in recruited patients
Overall survival | Five years
  Overall survival in recruited patients

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China